CLINICAL TRIAL: NCT02519218
Title: Outcomes Registry of Patients With Osteoarthritis and Varus Malalignment of the Knee Treated With Ellipse Intramedullary High Tibial Osteotomy (IM HTO) Nail System
Brief Title: Ellipse Intramedullary High Tibial Osteotomy Nail Study
Status: Completed | Type: Observational
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR0179
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis; Varus Malalignment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ellipse Technologies Intramedullary High Tibial Osteotomy Nail System

SUMMARY:
The purpose of this study is to collect outcomes data in patients implanted with the Ellipse IM HTO Nail System.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with the Ellipse IM HTO Nail System for osteoarthritis and varus malalignment of the knee
* Patient signs informed consent for the use of their personal private data.

Exclusion Criteria:

* Patient is currently enrolled in another clinical trial for high tibial osteotomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with the Ellipse IM HTO Nail system for osteoarthritis and varus malalignment of the knee.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Target vs. Actual Correction | Participants will be followed for the duration of correcting their deformity, an average of 3 weeks
  Measured as either weight-bearing line (percent) or HKA angle (degrees)
Target vs. Actual Correction | Participants will be followed for the duration of consolidation (bone healing), an average of 4 months
  Measured as either weight-bearing line (percent) or HKA angle (degrees)

SECONDARY OUTCOMES:
Change in Weight-Bearing Line | Participants will be followed for the duration of correcting their deformity, an average of 3 weeks
  Measured in percent
Change in Weight-Bearing Line | Participants will be followed for the duration of consolidation (bone healing), an average of 4 months
  Measured in percent
Change in Weight-Bearing Line | 1-year post-operative
  Measured in percent
Change in Weight-Bearing Line | 2-years post-operative
  Measured in percent
Change in Hip-Knee-Ankle Angle | Participants will be followed for the duration of correcting their deformity, an average of 3 weeks
  Measured in degrees
Change in Hip-Knee-Ankle Angle | Participants will be followed for the duration of consolidation (bone healing), an average of 4 months
  Measured in degrees
Change in Hip-Knee-Ankle Angle | 1-year post-operative
  Measured in degrees
Change in Hip-Knee-Ankle Angle | 2-years post-operative
  Measured in degrees
Change in Tibial Slope | Participants will be followed for the duration of correcting their deformity, an average of 3 weeks
  Measured in degrees
Change in Tibial Slope | Participants will be followed for the duration of consolidation (bone healing), an average of 4 months
  Measured in degrees
Change in Tibial Slope | 1-year post-operative
  Measured in degrees
Change in Tibial Slope | 2 years post-operative
  Measured in degrees
Time to full weight-bearing | Participants will be followed through 2 years post-operative
  Measured in days
Bone Healing | Participants will be followed for the duration of correcting their deformity, an average of 3 weeks
  Graded 0 through 2, corresponding to Not Healing, Healing, and Healed
Bone Healing | Participants will be followed for the duration of consolidation (bone healing), an average of 4 months
  Graded 0 through 2, corresponding to Not Healing, Healing, and Healed
Bone Healing | 1-year post-operative
  Graded 0 through 2, corresponding to Not Healing, Healing, and Healed
Bone Healing | 2 years post-operative
  Graded 0 through 2, corresponding to Not Healing, Healing, and Healed

OTHER OUTCOMES:
All Serious Adverse Events (SAEs) and Unanticipated Adverse Device Effects (UADEs) | Participants will be followed through 2 years post-operative
All non-serious adverse events in the limb related to the device or study procedure. Study procedure includes implant procedure and correction lengthening procedure. | Participants will be followed through 2 years post-operative
Secondary surgical procedures | Participants will be followed through 2 years post-operative
Surgical complications | Participants will be followed through 2 years post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dahl, MD, Principal Investigator — University of Minnesota